CLINICAL TRIAL: NCT02512445
Title: Trauma Informed Guilt Reduction Therapy
Acronym: TrIGR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Veterans Medical Research Foundation (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency); Brown University (Other); Seattle Institute for Biomedical and Clinical Research (Other); White River Junction Veterans Affairs Medical Center (U.S. Federal Agency); San Diego Veterans Healthcare System (U.S. Federal Agency); Providence VA Medical Center (U.S. Federal Agency); National Center for PTSD (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 09054
Record Dates: First submitted 2015-07-27; First posted 2015-07-30 (Estimated); Results first posted 2025-05-09 (Actual); Last update posted 2025-05-09 (Actual); Status verified 2025-05

CONDITIONS: Guilt; Shame; Post-traumatic Stress Disorders
MeSH Terms: conditions — Stress Disorders, Post-Traumatic | interventions — Palliative Care

STUDY DESIGN:
Intervention Model Description: 188 enrollment goal for primary study
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Trauma Informed Guilt Reduction Therapy (Experimental): 6-session psychotherapy intervention
  Interventions: Behavioral: Trauma Informed Guilt Reduction Therapy
- Supportive Care Therapy (Active Comparator): 6-session psychotherapy intervention
  Interventions: Behavioral: Supportive Care Therapy

INTERVENTIONS:
Behavioral: Trauma Informed Guilt Reduction Therapy — Trauma focused therapy
  Arms: Trauma Informed Guilt Reduction Therapy
Behavioral: Supportive Care Therapy — Supportive therapy
  Arms: Supportive Care Therapy

SUMMARY:
The goal of this project is to determine if a 6-session psychotherapy intervention will help Veterans feel less deployment-related guilt and less distress related to their guilt. Half of the participants will receive the guilt focused intervention and half will receive a supportive intervention. A supplemental pilot study added in FY2021 will examine the intervention for pandemic-related guilt events.

ELIGIBILITY:
Inclusion Criteria:

* Participant Served in OEF/OIF/OND, has post-traumatic guilt related to deployment event (for pandemic supplement in 2021, has guilt related to pandemic event)

Exclusion Criteria:

* Moderate or severe cognitive impairment, acute suicidality, current severe substance use disorder, unmanaged psychosis or mania

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 145 (Actual)
Dates: Start 2015-10 (Actual); Primary Completion 2023-06 (Actual); Study Completion 2023-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sonya B. Norman, PhD, Principal Investigator — Veterans Medical Research Foundation; Christy Capone, PhD, Principal Investigator — Brown University
Locations (3):
- United States (3):
  - VA San Diego Healthcare System, San Diego, California
  - National Center for PTSD, Boston, Massachusetts
  - VA Providence Medical Center, Providence, Rhode Island

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] McCue ML, Capone CC, Wachen JS, Harle KM, Davis BC, Panza KE, Lyons M, Luciano MT, Shea MT, Haller M, Galovski TE, Schnurr PP, Norman SB. Addressing pandemic-related guilt and shame in U.S. military veterans: A pilot randomized controlled trial of trauma-informed guilt reduction and supportive care therapy. Psychol Trauma. 2025 Oct 23:10.1037/tra0002036. doi: 10.1037/tra0002036. Online ahead of print. PMID 41129362
- [Derived] Capone C, Norman SB, Haller M, Davis B, Shea MT, Browne K, Lang AJ, Schnurr PP, Golshan S, Afari N, Pittman J, Allard CB, Westendorf L. Trauma Informed Guilt Reduction (TrIGR) therapy for guilt, shame, and moral injury resulting from trauma: Rationale, design, and methodology of a two-site randomized controlled trial. Contemp Clin Trials. 2021 Feb;101:106251. doi: 10.1016/j.cct.2020.106251. Epub 2020 Dec 14. PMID 33326878

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Trauma Informed Guilt Reduction Therapy | Supportive Care Therapy
Started | 74 | 71
Completed | 48 | 50
Not Completed | 26 | 21

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Trauma Informed Guilt Reduction Therapy | Supportive Care Therapy | Total
Number analyzed (Participants) | 74 | 71 | 145
Age, Continuous [Mean (Standard Deviation); unit: years] | 38.0 (7.6) | 40.5 (8.5) | 39.2 (8.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 4 | 9
  Male | 69 | 67 | 136
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 17 | 15 | 32
  Not Hispanic or Latino | 49 | 44 | 93
  Unknown or Not Reported | 8 | 12 | 20
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 4 | 9 | 13
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 6 | 7 | 13
  White | 49 | 43 | 92
  More than one race | 6 | 2 | 8
  Unknown or Not Reported | 9 | 10 | 19
Region of Enrollment [Number; unit: participants]
  United States | 74 | 71 | 145

OUTCOME MEASURES:

1. Primary Outcome: Trauma Related Guilt Inventory - Guilt Severity
Description: Change in Trauma Related Guilt Inventory - Guilt Severity Subscale Min score = 0, max score = 4 (score = mean of all items in subscale) higher scores = greater trauma related guilt severity
Time Frame: baseline to 8 months
Population: full sample
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Trauma Informed Guilt Reduction Therapy | Supportive Care Therapy
Number analyzed (Participants) | 74 | 71
score on a scale
  baseline | 2.5 [2.3 to 2.7] | 2.5 [2.3 to 2.7]
  follow-up | 1.6 [1.4 to 1.8] | 2.2 [1.9 to 2.4]

2. Secondary Outcome: Change in Clinician Administered Posttraumatic Stress Disorder (PTSD) Scale - 5 (CAPS-5)
Description: min = 0, max = 80 higher scores = more severe PTSD
Time Frame: baseline to 8 months
Population: full sample
Measure: Number (95% Confidence Interval); unit: score on a scale
Arm/Group | Trauma Informed Guilt Reduction Therapy | Supportive Care Therapy
Number analyzed (Participants) | 74 | 71
score on a scale
  baseline | 38.2 [35.5 to 40.9] | 38.6 [35.9 to 41.4]
  follow-up | 23.3 [20.2 to 26.4] | 30.9 [27.9 to 34.0]

3. Secondary Outcome: Change in Patient Health Questionnaire - 9 (PHQ-9)
Description: The PHQ-9 measures severity of depression symptoms. Scores range 0 - 27 higher scores = more severe depression
Time Frame: baseline to 8 months
Population: full sample
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Trauma Informed Guilt Reduction Therapy | Supportive Care Therapy
Number analyzed (Participants) | 74 | 71
score on a scale
  baseline | 15.1 [13.6 to 16.6] | 14.4 [12.9 to 15.9]
  follow up | 9.8 [8.0 to 11.5] | 12.5 [10.8 to 14.2]

4. Secondary Outcome: Change in Internalized Shame Scale
Description: change in Internalized Shame Scale scores range 0 to 120 higher scores = greater internalized shame
Time Frame: baseline to 8-month follow-up
Population: full sample
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Trauma Informed Guilt Reduction Therapy | Supportive Care Therapy
Number analyzed (Participants) | 74 | 71
score on a scale
  baseline | 51.4 [46.3 to 56.6] | 49.6 [44.3 to 54.8]
  follow up | 37.4 [31.6 to 43.1] | 41.9 [36.1 to 47.7]

5. Secondary Outcome: Change in World Health Organization Quality of Life - Brief
Description: Change in World Health Organization Quality of Life - Brief - score range = 0-100 higher scores = better quality of life
Time Frame: baseline to 8 months
Population: full sample
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Trauma Informed Guilt Reduction Therapy | Supportive Care Therapy
Number analyzed (Participants) | 74 | 71
score on a scale
  baseline | 43.7 [40.5 to 46.9] | 44.5 [41.3 to 47.8]
  follow up | 48.3 [44.6 to 51.9] | 44.4 [40.7 to 48.0]

6. Secondary Outcome: Change in Brief Symptom Inventory-18
Description: Change in Brief Symptom Inventory-18, a measure of depression, anxiety, and somatic symptoms score range = 0 - 72 higher scores = greater distress
Time Frame: baseline to 8 months
Population: full sample
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Trauma Informed Guilt Reduction Therapy | Supportive Care Therapy
Number analyzed (Participants) | 74 | 71
score on a scale
  baseline | 53.1 [50.9 to 55.3] | 54.0 [51.7 to 56.3]
  post treatment | 47.3 [44.8 to 49.9] | 49.0 [46.5 to 51.6]

ADVERSE EVENTS:
Time Frame: 6 months
Description: did not differ
Arm/Group | Trauma Informed Guilt Reduction Therapy | Supportive Care Therapy
All-Cause Mortality (participants affected / at risk) | 1/74 | 0/71
Serious Adverse Events (participants affected / at risk) | 0/74 | 0/71
Other Adverse Events (participants affected / at risk) | 4/74 | 8/71
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Trauma Informed Guilt Reduction Therapy (N=74) | Supportive Care Therapy (N=71)
increased suicidal ideation (Psychiatric disorders) | 1 (1) | 5 (5)
needed medical detox (Psychiatric disorders) | 2 (2) | 2 (2)
Arrested (Psychiatric disorders) | 1 (1) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2014-11-14): https://cdn.clinicaltrials.gov/large-docs/45/NCT02512445/Prot_SAP_000.pdf